CLINICAL TRIAL: NCT05227742
Title: Exploratory Study of the Effects of Low-Dose Psilocybin on Sensory Processing, Neurophysiological Arousal, and Emotional Health
Brief Title: Exploratory Study of Low Dose Psilocybin
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Diamond Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Peter Hendricks, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300008551
Record Dates: First submitted 2022-01-13; First posted 2022-02-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Demoralization
Keywords: Psilocybin; Low dose; Demoralization
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (0 mg psilocybin) (Placebo Comparator): Participants in this arm will receive 0 mg of psilocybin once per week for 5 weeks.
  Interventions: Drug: Placebo
- 1 mg psilocybin (Experimental): Participants in this arm will receive 1 mg psilocybin once per week for 5 weeks.
  Interventions: Drug: Psilocybin
- 2.5 mg psilocybin (Experimental): Participants in this arm will receive 2.5 mg psilocybin once per week for 5 weeks.
  Interventions: Drug: Psilocybin
- 5 mg psilocybin (Experimental): Participants in this arm will receive 5 mg psilocybin once per week for 5 weeks.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive oral psilocybin once per week for 5 weeks.
  Arms: 1 mg psilocybin; 2.5 mg psilocybin; 5 mg psilocybin
Drug: Placebo — Participants will receive inert placebo once per week for 5 weeks.
  Arms: Placebo (0 mg psilocybin)

SUMMARY:
The purpose of the present study is to evaluate the feasibility, initial signals of efficacy, and potential mechanisms of action of "microdoses" of psilocybin (i.e., low doses of psilocybin that are not believed to produce mystical-type, transcendent, hallucinogenic, or other overtly salient subjective effects that limit functionality) in the treatment of moderate to severe demoralization (feelings of hopelessness and meaningless that frequently accompany medical illness and other life hardship).

DETAILED DESCRIPTION:
Individuals who call research staff will undergo an initial telephone screen that will determine eligibility.

Week 1: Baseline Intake Appointment. Those who are eligible to participate on the basis of the telephone screen and provide informed consent will then complete a standard demographic questionnaire, a detailed psychiatric interview, and provide a urine sample for confirmation of substance abstinence and pregnancy status. Participants will then be administered a detailed medical history interview and physical examination including EKG and blood panel.

Week 2: Orientation. Participants who are medically eligible to participate will be scheduled for a psychoeducational orientation session that further explains the rationale of the study, and summarizes the study logistics. Participants will complete a number of baseline questionnaires and neuropsychological assessments at this time.

Week 3: Drug administration #1. In a between-groups design, participants will be randomized to receive 0 mg, 1 mg, 2.5 mg, or 5 mg of psilocybin at five weekly 6-hour long drug administration sessions. Dose will remain constant for each participant at each drug administration session.

At Drug Administration #1 and all subsequent drug administration sessions, participants will complete visual analogue scale (VAS) questions drawn from different sources that include drug abuse liability measures. These VAS questions will be administered at drug administration baseline and every 30 minutes thereafter through the end of acute effects at 6-hrs post-baseline. Research staff will complete a number of observational assessments at similar intervals.

Blood pressure will be assessed at regular intervals via automatic blood pressure monitor (i.e., at baseline and at 30, 60, 90, 120, 180, 240, and 360 min post-baseline), and medication for the treatment of acute hypertension will be administered should blood pressure exceed 200 systolic and/or 110 diastolic.

At peak drug effects (2 hr post-baseline), a number of measures will be administered, each differing by drug administration session. At Drug Administration #1, participants will undergo two electroencephalogram (EEG) tasks (with assessments at baseline serving as pre-drug control values).

At 6-hr post-baseline, participants will complete self-report measures assessing the subjective experience. These questionnaires will be administered at the conclusion of each drug administration session. Participants will then be administered a brief semi-structured qualitative interview designed to probe the nature of their experience. All participants will be required to arrange for transportation home from the CRU; participants will not be allowed to drive themselves after drug administration sessions.

Week 4: Drug Administration #2. This session will be identical to Drug Administration #1, however, at peak drug effects, participants will complete two new EEG tasks (with assessments at baseline serving as pre-drug control values).

Week 5: Drug Administration #3. This session will be identical to prior drug administration sessions, however, at peak drug effects, a neuropsychological measure will be administered.

Week 6: Drug Administration #4. This session will be identical to prior drug administration sessions, however, at peak drug effects, participants will complete another neuropsychological measure.

Week 7: Drug Administration #5. This session will be identical to prior drug administration sessions, however, at peak drug effects, participants will complete another neuropsychological measure. At the conclusion of this measure, subjects will undergo an EEG assessment (with an assessment at baseline serving as a pre-drug control value).

Week 8: Study Termination. This session will comprise completion of the same questionnaires that were previously completed at baseline as well as a semi-structured qualitative interview. EKG will be repeated at study termination.

It is noted that over the duration of the study, every day participants will be asked to complete some brief self-report measures and a resting state EEG via a smartphone app.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read and write in English
2. Between 25 and 65 years old
3. Demoralization Scale-II (DS-II) score of > 8
4. No prior hallucinogen use or it would have been 3 years since the last use of a hallucinogen
5. Availability of a friend, family member, or other form of transportation (e.g., Uber) to drive participants home after their drug administration sessions
6. In good general health as assessed by detailed medical history interview and physical examination

Exclusion Criteria:

1. 24 years of age or younger; 66 years of age or older
2. Women who are pregnant (pregnancy status confirmed via urine pregnancy test) or breastfeeding
3. Current hypertension (exceeding 140 systolic and/or 90 diastolic at resting)
4. Use of methylphenidate or other medications for ADHD, benzodiazepines or other medications for anxiety (e.g., beta-blockers), tricyclic antidepressants, MAOIs, SSRIs, SNRIs or other medications for depression, lithium or other mood stabilizers, haloperidol or other antipsychotic medications, any medications or supplements with serotonin activity (e.g., St. John's Wort), or any other pharmacologic or biologic agent used to treat depression or anxiety (e.g., magnesium, cannabis)
5. Personal or family history (first or second degree relatives) of psychotic or bipolar I or II disorders
6. Any suicidal ideation of type 4 or type 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) in the 3 months prior to screening (i.e., active suicidal thought with method and intent but without a specific plan, or active suicidal thought with method, intent and plan).
7. History of head trauma, loss of consciousness, or neurological disease
8. Receiving treatment within the past 30 days for depression, anxiety, or substance use disorder
9. Participation within the past 30 days in a clinical trial for the treatment of depression, anxiety, or substance use disorder
10. Any current substance use disorder diagnosis (substance abstinence confirmed via urine drug screen)
11. History of immoderate alcohol consumption within the past 3 months per NIAAA definitions: more than 4 drinks per day or 14 drinks per week for men; more than 3 drinks per day or 7 drinks per week for women
12. Any headache disorder (i.e., migraine, tension-type headache, or cluster headache) in the past year
13. Planning to move from the Birmingham area in the next 3 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Demoralization | Study Termination at Week 8
  Demoralization as assessed by the Demoralization Scale-II (DS-II; possible range = 0 to 32, with higher scores reflecting worse outcomes)
Mystical Experience | At the conclusion of Drug Administration #1 at Week 3
  Mystical experience as assessed by the Mystical Experience Questionnaire (MEQ; possible range = 0 to 5, with higher scores reflecting more mystical experience)
Mystical Experience | At the conclusion of Drug Administration #2 at Week 4
  Mystical experience as assessed by the Mystical Experience Questionnaire (MEQ; possible range = 0 to 5, with higher scores reflecting more mystical experience)
Mystical Experience | At the conclusion of Drug Administration #3 at Week 5
  Mystical experience as assessed by the Mystical Experience Questionnaire (MEQ; possible range = 0 to 5, with higher scores reflecting more mystical experience)
Mystical Experience | At the conclusion of Drug Administration #4 at Week 6
  Mystical experience as assessed by the Mystical Experience Questionnaire (MEQ; possible range = 0 to 5, with higher scores reflecting more mystical experience)
Mystical Experience | At the conclusion of Drug Administration #5 at Week 7
  Mystical experience as assessed by the Mystical Experience Questionnaire (MEQ; possible range = 0 to 5, with higher scores reflecting more mystical experience)
Challenging Experience | At the conclusion of Drug Administration #1 at Week 3
  Challenging experience as assessed by the Challenging Experience Questionnaire (CEQ; possible range = 0=5, with higher scores reflection more challenging experiences)
Challenging Experience | At the conclusion of Drug Administration #2 at Week 4
  Challenging experience as assessed by the Challenging Experience Questionnaire (CEQ; possible range = 0=5, with higher scores reflection more challenging experiences)
Challenging Experience | At the conclusion of Drug Administration #3 at Week 5
  Challenging experience as assessed by the Challenging Experience Questionnaire (CEQ; possible range = 0=5, with higher scores reflection more challenging experiences)
Challenging Experience | At the conclusion of Drug Administration #4 at Week 6
  Challenging experience as assessed by the Challenging Experience Questionnaire (CEQ; possible range = 0=5, with higher scores reflection more challenging experiences)
Challenging Experience | At the conclusion of Drug Administration #5 at Week 7
  Challenging experience as assessed by the Challenging Experience Questionnaire (CEQ; possible range = 0=5, with higher scores reflection more challenging experiences)
PASAT | At hour 2 of Drug Administration #3 at Week 5
  Executive functioning as assessed by the Paced Auditory Serial Addition Test (PASAT)
Trail Making | At hour 2 of Drug Administration #4 at Week 6
  Executive functioning as assessed by the Delis-Kaplan Trail Making Test
CPT-3 | At hour 2 of Drug Administration #5 at Week 7
  Attention and cognitive control as assessed by Conner's Continuous Performance Test (CPT-3)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States